CLINICAL TRIAL: NCT03414268
Title: A Phase 3, Prospective, Double-Blinded, Randomized Controlled Trial of the Micronized dHACM Injection As Compared To Saline Placebo Injection In The Treatment Of Plantar Fasciitis
Brief Title: Micronized dHACM Injectable for the Treatment of Plantar Fasciitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MiMedx Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AIPF007
Record Dates: First submitted 2018-01-23; First posted 2018-01-29 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2020-10

CONDITIONS: Fasciitis, Plantar
Keywords: Chronic plantar fasciitis; Heel pain
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Micronized dHACM (Experimental): 1 mL injection of 40 mg Micronized dehydrated human amnion/chorion membrane (dHACM)
  Interventions: Other: Micronized dHACM
- Saline Injection (Placebo Comparator): Injection of 1mL 0.9% Sodium Chloride Injection, USP
  Interventions: Drug: Saline Injection

INTERVENTIONS:
Other: Micronized dHACM — 1 mL injection of 40 mg Micronized dehydrated human amnion/chorion membrane (dHACM)
  Other Names: dHACM
  Arms: Micronized dHACM
Drug: Saline Injection — Injection of 1mL 0.9% Sodium Chloride Injection, USP
  Other Names: 0.9% NaCl; Normal Saline; Sodium Chloride Injection, USP
  Arms: Saline Injection

SUMMARY:
Prospective, double-blinded, randomized controlled trial of the micronized dHACM injection as compared to the saline placebo injection in the treatment of plantar fasciitis

DETAILED DESCRIPTION:
Approximately 276 patients will be enrolled in this study. Each patient will receive 1 injection and be evaluated for efficacy and safety during a 6-month observation period. Randomization will be 1:1. The study is expected to be completed within 34 months, inclusive of enrollment and follow-up of all subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of plantar fasciitis for ≥ 1 month (30 days) and ≤ 18 months by the investigator
2. VAS Pain scale of ≥ 45 mm at randomization
3. Plantar fasciitis with conservative treatment for ≥ 1 month (30 days), including any of the following modalities:

   * RICE
   * Stretching exercises
   * NSAIDs
   * Orthotics
4. Diagnostic X-Ray within 6 months of enrollment showing view of calcaneus negative for calcaneal fracture or structural abnormalities
5. BMI ≤ 40 kg/m2
6. Age ≥ 21 years and < 80 years
7. Ability to sign Informed Consent and Release of Medical Information Forms
8. Ability to receive and respond to text messages or emails on a daily basis.

Exclusion Criteria:

1. Prior surgery or trauma to the affected site
2. Subjects requiring bilateral plantar fasciitis treatment at time of enrollment
3. Prior use of any lower limb injection therapy, including corticosteroids or PRP in either limb within the last 3 months
4. Has diabetes either Type I or Type II.
5. Systemic disorders associated with enthesopathy (disorder of entheses, i.e. bone attachments) such as Gout, Reiter's syndrome, rheumatoid arthritis, etc.
6. The presence of diagnosed comorbidities that can be confused with or can exacerbate the condition- to be assessed by X-ray - including but not limited to:

   * Calcaneal stress fracture
   * Nerve entrapment syndrome (diagnosed as Baxter Nerve Syndrome)
   * Fat pad atrophy
   * Acute traumatic rupture of the plantar fascia
   * Calcaneal tumor
   * Tarsal tunnel syndrome (diagnosed)
   * Significant bone deformity of the foot that may interfere with the study
7. Affected site exhibits clinical signs and symptoms of infection
8. Known allergy or known sensitivity to Aminoglycosides
9. Subjects who are non-ambulatory
10. History of more than 14 days treatment with immuno-suppressants (including systemic corticosteroids) or cytotoxic chemotherapy within 30 days prior to enrollment, or who are anticipated to require such medications during the course of the study
11. Prior radiation at the site
12. Use of any investigational drug(s) or therapeutic device(s) within 3 months preceding enrollment
13. Immune disorders including Systemic Lupus Erythematosus (SLE), Fibromyalgia, Acquired Immunodeficiency Syndrome (AIDS) or Human Immunodeficiency Virus (HIV)
14. History of any condition (including drug or alcohol abuse, medical or psychiatric condition) that is likely to impair understanding of or compliance with the study protocol, in the judgment of the investigator
15. Pregnancy at enrollment or within last 6 months, women who are breastfeeding, or women of childbearing potential who are planning to become pregnant during the time of the study OR are unwilling/unable to use acceptable methods of contraception (birth control pills, barriers, or abstinence)
16. Workers' compensation subjects

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2021-03-17 (Actual); Study Completion 2021-03-17 (Actual)

PRIMARY OUTCOMES:
Change in VAS score | 90 Days
  Visual Analog Scale for Pain:
Incidence of adverse events | 180 Days
  The incidence of related Adverse Events (AEs), Serious Adverse Events (SAEs), and Unanticipated Adverse Events during the first 12 months post injection

SECONDARY OUTCOMES:
Foot Function Index - Revised (FFI-R) (Short Form) | 90 Days
  Foot Function Index - Revised: Patient Reported Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Stuart D Miller, MD, Principal Investigator — MedStar Union Memorial Hospital, Baltimore, MD
Locations (17):
- United States (17):
  - Southern Arizona VA Health Care System, Tucson, Arizona
  - ILD Research Center, Carlsbad, California
  - Center for Clinical Research, Carmichael, California
  - Limb Preservation Platform, Inc., Fresno, California
  - Horizon Clinical Research, La Mesa, California
  - Foot and Ankle Clinic, Los Angeles, California
  - Five Cities Foot Clinic, Pismo Beach, California
  - Bay Pines VA Healthcare System, Bay Pines, Florida
  - Gulfcoast Research Institute, LLC, Sarasota, Florida
  - Doctors Research Network, South Miami, Florida
  - Union Podiatry, Baltimore, Maryland
  - Advanced Foot & Ankle Center, Las Vegas, Nevada
  - University Orthopedics Center, Altoona, Pennsylvania
  - University Orthopedics Center, State College, Pennsylvania
  - Futuro Clinical Trials, LLC, McAllen, Texas
  - Endeavor Clinical Trials, San Antonio, Texas
  - Coastal Podiatry, Virginia Beach, Virginia